CLINICAL TRIAL: NCT06281925
Title: A Phase II Randomized Interventional Pilot Study for Colon Cancer Patients Receiving Oxaliplatin: Benefits of Cryotherapy in Prevention of Peripheral Neuropathy
Brief Title: Cryotherapy & Oxaliplatin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01363
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer; Peripheral Neuropathy
MeSH Terms: conditions — Colonic Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryotherapy (Experimental): Patients receiving oxaliplatin who are randomized to the Interventional (Cryotherapy) Arm will wear a pair of gloves that has removable ice packs throughout their treatment, starting 15 minutes before and ending 15 minutes after completion of oxaliplatin. These ice packs will be replaced every 30 minutes. The total wearing time of the cryotherapy will be approximately 2 hours.
  Interventions: Device: Cryotherapy Gloves
- Control (No Intervention): Patients receiving oxaliplatin who are randomized to the Control Arm will not receive the gloves with removable ice packs throughout their treatment.

INTERVENTIONS:
Device: Cryotherapy Gloves — All patients in the intervention group will receive cryotherapy with cold packs enclosed in a fabric envelope (gloves). The fabric envelope (gloves) will be patient specific.
  Arms: Cryotherapy

SUMMARY:
The primary objective of this study is to determine if cryotherapy is beneficial to patients with colon cancer who are receiving oxaliplatin in the prevention of developing chemotherapy induced peripheral neuropathy.

DETAILED DESCRIPTION:
Peripheral neuropathy often manifests as numbness and tingling in the hands and feet, which may be detrimental to the patients' overall safety and quality of life, thereby causing them to stop or delay treatment. Everyday tasks such as walking, buttoning a shirt, or tying shoes can become challenging. Select chemotherapy agents are known to cause significant peripheral neuropathy. Studies have been performed demonstrating efficacy of using cryotherapy, which causes vasoconstriction, to targeted areas of the body, in relation to paclitaxel. These studies have shown drastic differences between those who receive cryotherapy during treatment and those who do not. There are few studies on the use of cryotherapy in the prevention of peripheral neuropathy with the use of oxaliplatin, which will be undertaken in this study.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Willingness to participate in research
* Diagnosed with stage III colon cancer
* Chemotherapy naïve
* Planning to initiate Capecitabine + Oxaliplatin (CAPOX) chemotherapy regimen as part of standard of care.

Exclusion Criteria:

* Pre-existing peripheral neuropathy
* Pre-existing diabetes
* Raynaud's disease
* Metabolic syndrome, including: Hypertension; Hypercholesterolemia; and Obesity (BSA > 2)
* Upper extremity amputees
* Specific autoimmune diseases: Guillain-Barre; Lupus; Rheumatoid arthritis; and Sjogren's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Peripheral Neuropathy at Visit 2 | Visit 2 (Day 1)
  Presence of peripheral neuropathy will be evaluated using common terminology criteria for adverse events (CTCAE) version 5.
Proportion of Participants with Peripheral Neuropathy at Visit 3 | Visit 3 (Day 21)
  Presence of peripheral neuropathy will be evaluated using common terminology criteria for adverse events (CTCAE) version 5.
Proportion of Participants with Peripheral Neuropathy at Visit 4 | Visit 4 (Day 42)
  Presence of peripheral neuropathy will be evaluated using common terminology criteria for adverse events (CTCAE) version 5.
Proportion of Participants with Peripheral Neuropathy at Visit 5 | Visit 5 (Day 63)
  Presence of peripheral neuropathy will be evaluated using common terminology criteria for adverse events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mendez, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, Mineola, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: sarah.mendez@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to sarah.mendez@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.